CLINICAL TRIAL: NCT03699033
Title: A Phase II Trial of Hypofractionated Intensity-Modulated Radiation Therapy (IMRT) Utilizing 2.5 Gy/Fraction to PET-avid Disease Combined With Carboplatin and Paclitaxel for Subjects With Stage IIIA or IIIB Non-Small Cell Lung Cancer
Brief Title: Hypofractionated Radiotherapy With Carboplatin and Paclitaxel in Non-Small Cell Lung Cancer
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: No patients available
Sponsor: Stephanie Smiddy (Other)
Responsible Party: Sponsor-Investigator, Stephanie Smiddy, Investigator, University of Toledo Health Science Campus
Organization: University of Toledo (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 202923
Record Dates: First submitted 2018-10-03; First posted 2018-10-09 (Actual); Last update posted 2020-11-05 (Actual); Status verified 2018-10

CONDITIONS: Non Small Cell Lung Cancer
Keywords: Radiation; NSCLC; Hypofractionated; Carboplatin; Paclitaxel; IMRT; Fraction; Stage III; 4D PET/CT
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Carboplatin; Paclitaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Radiation (Experimental): 2.5 Gy/Fraction
  Interventions: Radiation: 2.5 Gy/fraction; Drug: Carboplatin; Drug: Paclitaxel

INTERVENTIONS:
Radiation: 2.5 Gy/fraction — Hypofractionated Intensity-Modulated Radiation Therapy (IMRT) Utilizing 2.5 Gy/Fraction to PET-avid Disease Combined with Carboplatin and Paclitaxel
Drug: Carboplatin — The doses of chemotherapy to be given concurrently with conformal radiotherapy will be weekly paclitaxel (45 mg/m2) and carboplatin (AUC=2), respectively.
  Consolidation chemotherapy with 2 cycles of carboplatin (AUC=6) and paclitaxel (200 mg/m2) should be administered following completion of concurrent chemoradiation.
Drug: Paclitaxel — The doses of chemotherapy to be given concurrently with conformal radiotherapy will be weekly paclitaxel (45 mg/m2) and carboplatin (AUC=2), respectively.
  Consolidation chemotherapy with 2 cycles of carboplatin (AUC=6) and paclitaxel (200 mg/m2) should be administered following completion of concurrent chemoradiation.

SUMMARY:
Single center, single arm, Phase II study designed to evaluate the feasibility of hypofractionated IMRT to 62.5 Gy in 25 fractions (2.5 Gy/fraction) with 4D PET/CT-based radiation treatment planning and concurrent carboplatin and paclitaxel in Stage IIIA or Stage IIIB NSCLC subjects.

DETAILED DESCRIPTION:
This study is designed to evaluate the feasibility of hypofractionated IMRT to 62.5 Gy in 25 fractions (2.5 Gy/fraction) with 4D PET/CT-based radiation treatment planning and concurrent carboplatin and paclitaxel in Stage IIIA or Stage IIIB NSCLC subjects.

Hypofractionated IMRT allows escalation of the biological effective dose (BED) to the tumor and reduces the radiation treatment duration to 5 weeks. Increasing the BED without protracting the RT course may be a more effective means of dose escalation than simply increasing the total dose but using only 2 Gy/fraction, as was tested in RTOG 0617.

Investigators require the use of advanced treatment planning techniques, including 4D CT simulation, volume delineation utilizing PET/CT to identify gross disease and IMRT to minimize the total volume of normal tissue receiving a high dose of radiation.

As minimal published work has evaluated hypofractionated RT regimens for Stage III NSCLC with concurrent chemotherapy, investigators selected a moderately escalated dose/fraction of 2.5 Gy for evaluation in combination with concurrent carboplatin and paclitaxel.

ELIGIBILITY:
Inclusion Criteria:

* Pathologically proven diagnosis of Stage IIIA or IIIB non-small cell lung cancer (NSCLC).
* Stage IIIA subjects who are considered eligible for resection following neoadjuvant chemoradiation are eligible for this study.
* No PET/CT evidence of metastatic disease.
* An MRI of the brain with contrast excluding intracranial metastatic disease (or CT with contrast if MRI is medically contraindicated). An MRI without contrast is only permitted if the subject cannot have contrast for medical reasons.
* If a pleural effusion is present, it must be tapped and confirmed to be cytologically negative. If an effusion is deemed too small to safely tap, the subject will be eligible.
* Subjects must have measurable or evaluable disease.
* No prior thoracic radiotherapy.
* Age > 18 years at time of registration.
* ECOG Performance Status of 0-2 (Karnofsky performance scale ≥ 60).
* Hgb > 9 g/dL; ANC (absolute neutrophil count) > 1500/µl; platelets > 100,000 mcL.
* Subjects must sign study-specific informed consent form prior to registration.
* Radiation therapy and chemotherapy must start within 4 weeks of study enrollment.

Exclusion Criteria:

* Evidence of severe or uncontrolled psychiatric or systemic disease (e.g., unstable or uncompensated respiratory, cardiac, hepatic, or renal disease) that would interfere with study protocol as judged by the investigator.
* Active connective tissue disorders, such as active lupus or scleroderma.
* Known Acquired Immune Deficiency (HIV (+)/AIDS).
* Subjects must not be pregnant or nursing due to the potential for congenital abnormalities and the potential of this regiment to harm nursing infants. Women of childbearing potential must agree to use medically approved and adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry, for the duration of study participation, and for 90 days following completion of therapy. Should a woman become pregnant or suspect she is pregnant while participating in this study, she should inform her treating physician immediately.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2018-10-01 (Actual); Primary Completion 2020-10-01 (Actual); Study Completion 2020-10-01 (Actual)

PRIMARY OUTCOMES:
Acute and late toxicities assessed based on the common toxicity criteria for adverse events version 3.0 (CTCAEv5.0) | During and within 90 days of radiation therapy
  Acute toxicities (toxicity during and within 90 days of radiation therapy) and delayed toxicities will be measured using CTCAE criteria, version 5.0. Acute toxicities are defined as those toxicities occurring during and within 90 days from the completion of radiotherapy and delayed toxicities are those that develop at least 90 days after the last dose of radiation

SECONDARY OUTCOMES:
Progression-free survival | year 0 - year 2
  Progression-free survival will be measured from the last day of radiation treatment until evidence of local or distant disease progression.
Overall Survival | year 0 - year 5
  Overall survival will be measured from the last day of radiation treatment until death.
Local control | year 0 - year 2
  Assessment of local control after treatment with radiotherapy combined with Carboplatin and Placlitaxel

CONTACTS AND LOCATIONS:
Locations (1):
- University of Toledo, Eleanor N. Dana Cancer Center, Toledo, Ohio, United States

IPD SHARING:
Plan to Share IPD: Undecided